CLINICAL TRIAL: NCT01206465
Title: A Phase I Clinical Trial of Sequential Pralatrexate Followed by a 48-hour Infusion of 5- Fluorouracil Given Every Other Week in Adult Patients With Solid Tumors
Brief Title: Pralatrexate and Fluorouracil in Treating Patients With Recurrent Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0238-10-FB; NCI-14191 (Other Grant/Funding Number: National Cancer Institute)
Record Dates: First submitted 2010-09-17; First posted 2010-09-21 (Estimated); Results first posted 2018-07-16 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: interventions — 10-propargyl-10-deazaaminopterin; Fluorouracil; Chromatography, High Pressure Liquid; Polymerase Chain Reaction; Base Sequence; Pharmacogenomic Testing; Amplified Fragment Length Polymorphism Analysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (enzyme inhibitor therapy) (Experimental): Patients receive pralatrexate IV over 5 minutes on day 1 and fluorouracil IV continuously over 48 hours on days 2 and 16. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: pralatrexate; Drug: fluorouracil; Other: laboratory biomarker analysis; Genetic: DNA analysis; Other: high performance liquid chromatography; Genetic: polymerase chain reaction; Genetic: nucleic acid sequencing; Other: pharmacological study; Other: pharmacogenomic studies; Genetic: polymorphism analysis

INTERVENTIONS:
Drug: pralatrexate — Given IV
  Other Names: FOLOTYN; PDX
Drug: fluorouracil — Given IV
  Other Names: 5-fluorouracil; 5-Fluracil; 5-FU
Other: laboratory biomarker analysis — Correlative studies
Genetic: DNA analysis — Correlative studies
Other: high performance liquid chromatography — Correlative studies
  Other Names: HPLC
Genetic: polymerase chain reaction — Correlative studies
  Other Names: PCR
Genetic: nucleic acid sequencing — Correlative studies
  Other Names: Gene Sequencing; Molecular Biology, Nucleic Acid Sequencing
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: pharmacogenomic studies — Correlative studies
  Other Names: Pharmacogenomic Study
Genetic: polymorphism analysis — Correlative studies

SUMMARY:
RATIONALE: Pralatrexate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as fluorouracil, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving pralatrexate together with fluorouracil may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of pralatrexate when given together with fluorouracil in treating patients with recurrent solid tumors

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the recommended dose of PDX (pralatrexate) given in combination with a fixed dose of 5-FU (fluorouracil) administered as a 48-hour infusion given every other week.

SECONDARY OBJECTIVES:

I. To assess clinical response to therapy in subjects with measurable disease and time to disease progression in all subjects.

II. To assess the toxicity profile of the combination of PDX and 5-FU. III. To determine the pharmacokinetics of PDX and 5-FU and correlate with clinical toxicity.

IV. To analyze polymorphisms in methylenetetrahydrofolate reductase and thymidylate synthase (TS) and correlate with clinical toxicity.

OUTLINE: This is a dose-escalation study of pralatrexate.

Patients receive pralatrexate intravenously (IV) over 5 minutes on day 1 and fluorouracil IV continuously over 48 hours on days 2 and 16. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Cancer patients who have failed standard therapy for their disease or for whom no such therapy is available are eligible, for which 5-fluoropyrimdines, including 5-FU, or inhibitors of DHFR (dihydrofolate reductase), including pralatrexate, have the potential for therapeutic benefit
* Objectively measurable disease is preferred, but not required
* Performance status of 0-2 (Eastern Cooperative Oncology Group [ECOG])
* Prior treatment:
* The patient should have recovered from the toxicities associated with prior chemotherapy (at least 3 weeks from prior therapy)
* At least two or more weeks should have elapsed since any radiotherapy, and the patient should have recovered from the toxicity associated with such therapy
* If a recent surgical procedure has been performed, the patient should have recovered from the surgery prior to entering this trial
* Absolute granulocyte count of 1500 per mcL or greater
* Platelet count of 100,000 per mcL or greater
* Serum bilirubin less than 1.5 times the upper limits of the institutional normal
* Serum creatinine less than the upper limits of normal
* The patient must willingly give signed informed consent

Exclusion Criteria:

* Pregnant women and nursing mothers are ineligible; eligible patients of reproductive potential should use adequate contraception if sexually active
* Serious concurrent medical illness which would jeopardize the ability of the patient to receive the chemotherapy program outlined in this protocol with reasonable safety
* Patients with active infections requiring intravenous antibiotic therapy are not eligible until the infection has resolved
* Patients who are human immunodeficiency virus (HIV) antibody positive and are receiving highly active antiretroviral therapy (HAART) are ineligible
* Concomitant administration of nonsteroidal anti-inflammatory drugs (NSAIDs) and trimethoprim/sulfamethoxazole will not be allowed

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2010-09-14 (Actual); Primary Completion 2015-02-04 (Actual); Study Completion 2017-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean Grem, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Eppley Cancer Center, Omaha, Nebraska, United States

REFERENCES:
- [Result] Grem JL, Kos ME, Evande RE, Meza JL, Schwarz JK. A phase 1 clinical trial of sequential pralatrexate followed by a 48-hour infusion of 5-fluorouracil given every other week in adult patients with solid tumors. Cancer. 2015 Nov 1;121(21):3862-8. doi: 10.1002/cncr.29504. Epub 2015 Aug 4. PMID 26242208

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 29 signed a consent form. Two patients never received any study drug: one became ineligible due to rise in bilirubin; another decided against participating.
Groups:
- 75 mg/m^2; 94 mg/m^2; 118 mg/m^2; 148 mg/m^2; 185 mg/m^2: pralatrexate (PDX) dose level
Period: Overall Study
Arm/Group | 75 mg/m^2 | 94 mg/m^2 | 118 mg/m^2 | 148 mg/m^2 | 185 mg/m^2
Started | 3 | 6 | 6 | 6 | 6
Completed | 3 | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis was performed on 27 patients who received study drug; 2 patients did not receive any study drug (1 changed mind after signing consent; 1 no longer eligible due to elevated bilirubin)
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 27
Age, Continuous [Median (Full Range); unit: years] | 61 [30 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 14
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Caucasian | 24
  Race/Ethnicity: Black, not of hispanic origin | 1
  Race/Ethnicity: Hispanic | 1
  Race/Ethnicity: Asian | 1
Region of Enrollment [Number; unit: participants]
  United States | 27

OUTCOME MEASURES:

1. Primary Outcome: Recommended Dose of PDX Given With a Fixed Dose of 5-FU
Description: Recommended dose of PDX given in combination with a fixed dose of 5-FU administered as a 48-hour infusion given every other weekMaximum tolerated dose will have been exceeded when 2 patients entered at a given dose level experience specified dose-limiting toxicities in the initial cycle
Time Frame: During the initial course (day 1 & 15 of a 4 week schedule)
Population: All participants receive pralatrexate IV over 5 minutes on day 1 and fluorouracil IV continuously over 48 hours on days 2 and 16. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
Measure: Number; unit: mg per meter square
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 27
mg per meter square | 148

2. Secondary Outcome: Response to Therapy in Subjects With Measurable Disease
Description: Number of Participants With Response to Therapy in Subjects With Measurable Disease
Time Frame: restaging imaging done after each two 4-week course until time of progression (the maximum duration of PFS = 588 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 27
Participants
  complete or partial response | 0
  stable disease | 18
  progressive disease | 9

3. Secondary Outcome: Number of Patients Experiencing Grade 3-4 Toxicity While Receiving the Combination of PDX and 5-FU
Description: Participants remained on study as long as they did not progress, and wished to continue on study (no limit on number of cycles)
Time Frame: ., "From the time the subject signs the consent form and ending 4 weeks following the final chemotherapy, an average of 3 years
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 27
participants
  gr 3-4 neutropenia | 4
  gr 3-4 thrombocytopenia | 0
  gr 3-4 anemia | 4
  gr 3-4 diarrhea | 1
  gr 3-4 mucositis | 5
  gr 3-4 dehydration | 1
  gr 3-4 fatigue | 1

4. Secondary Outcome: Pharmacokinetics of PDX- AUClast
Description: Plasma concentrations versus time (at all time points)
Time Frame: Pre-treatment, end of infusion, at 15, 30, and 60 min, and then at 2, 4, 6, 8, 12, 22, 23, 24, 45, and 46 hours for PDX.
Population: AUClast
Measure: Mean (Standard Deviation); unit: ng/ml *hr
Groups:
- 75 mg/m^2: pralatrexate (PDX) Dose level 1
- 94 mg/m^2: PDX Dose Level 2
- 118 mg/m^2: PDX Dose level 3
- 148 mg/m^2: PDX Dose level 4
- 185 mg/m^2: PDX Dose level 5
Arm/Group | 75 mg/m^2 | 94 mg/m^2 | 118 mg/m^2 | 148 mg/m^2 | 185 mg/m^2
Number analyzed (Participants) | 3 | 6 | 6 | 6 | 6
ng/ml *hr | 12,818 (578) | 16300 (728) | 15680 (801) | 23570 (2411) | 42121 (1051)

5. Secondary Outcome: Polymorphisms in Methylenetetrahydrofolate Reductase and Thymidylate Synthase
Description: Number of Participants with Polymorphisms in Methylenetetrahydrofolate Reductase and Thymidylate Synthase
Time Frame: Prior to the first dose of protocol therapy
Measure: Number; unit: percentage of patients
Groups:
- Wild Type: The phenotype generally found in a natural population
- Heterozygous: Different alleles or versions of a gene
- Homozygous Variant: Same alleles or versions of a gene
Arm/Group | Wild Type | Heterozygous | Homozygous Variant
Number analyzed (Participants) | 27 | 27 | 27
percentage of patients
  SLC19A1 80G>A | 51.9 | 40.7 | 7.4
  gamma glutamyl hydrolase (GGH) 401C>T | 55.6 | 37.0 | 7.4
  gamma glutamyl hydrolase (GGH) 452C>T | 88.9 | 11.1 | 0
  folyl polyglutamate synthase (FPGS) rs10760502A>G | 96.0 | 4.0 | 0
  folyl polyglutamate synthase (FPGS) rs1544105C>T | 25.9 | 55.6 | 18.5
  methylene tetrahydrofolate reductase (MTHFR 677C>T | 55.6 | 25.9 | 18.5
  methylene tetrahydrofolate reductase MTHFR 1298A>C | 51.9 | 33.3 | 14.8
  thymidylate synthase 28-bp tandem repeats (2 or 3) | 14.8 | 48.2 | 37.0

6. Secondary Outcome: 5-FU Plasma Levels
Description: Pharmacokinetics of 5-FU - Cmax plasma levels
Time Frame: 22, 23, 45 & 46 hours during the 48 hour infusion
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/m^2
Groups:
- 22 Hours; 23 Hours; 45 Hours; 46 Hours: 5 FU plasma levels
Arm/Group | 22 Hours | 23 Hours | 45 Hours | 46 Hours
Number analyzed (Participants) | 27 | 27 | 27 | 27
mg/m^2 | 1147 (133) | 1159 (121) | 1123 (130) | 1113 (135)

7. Secondary Outcome: Time to Disease Progression
Description: Time to disease progression in all Participants
Time Frame: restaging imaging done after each two 4-week course until time of progression (longest time to progression = 588 days)
Population: as for outcome 1
Measure: Median (Full Range); unit: days
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 27
days | 112 [28 to 588]

ADVERSE EVENTS:
Time Frame: Adverse event data is collected on participants from the time of consent until 30 days after the participant is off study drug.
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
All-Cause Mortality (participants affected / at risk) | 3/27
Serious Adverse Events (participants affected / at risk) | 10/27
Other Adverse Events (participants affected / at risk) | 27/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Enzyme Inhibitor Therapy) (N=27)
Thromboembolic Event (Vascular disorders) | 4 (4) — Pulmonary emboli
Pain (General disorders) | 2 (2)
gastrointestinal disorders - Other (Gastrointestinal disorders) | 1 (1) — diverticulitis
Nervous system disorders- Other (Nervous system disorders) | 1 (1) — mental status change
Sepsis (Infections and infestations) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (3)
Fracture (Injury, poisoning and procedural complications) | 1 (1) — tibia bone
Wound complication (Injury, poisoning and procedural complications) | 1 (2) — surgery
hypotension (Vascular disorders) | 1 (1)
Infection and infestations- Other (Infections and infestations) | 1 (1) — related to mucositis
Joint infection (Infections and infestations) | 1 (1) — knee
Diarrhea (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Enzyme Inhibitor Therapy) (N=27)
Hemoglobinuria (Renal and urinary disorders) | 5 (10)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (2)
Mucositis oral (Gastrointestinal disorders) | 23 (23)
Ascites (Gastrointestinal disorders) | 2 (2)
white blood cell decreased (Investigations) | 2 (3)
Localized Edema (General disorders) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2)
Neutrophil count decreased (Investigations) | 13 (13)
Platelet count decreased (Investigations) | 16 (16)
Anemia (Blood and lymphatic system disorders) | 20 (20)
Diarrhea (Gastrointestinal disorders) | 11 (11)
dehydration (Metabolism and nutrition disorders) | 9 (9)
Fatigue (General disorders) | 15 (15)
rash, maculo-papular (Skin and subcutaneous tissue disorders) | 7 (7)
Nausea (Gastrointestinal disorders) | 8 (8)
constipation (Gastrointestinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No